CLINICAL TRIAL: NCT02335359
Title: Tranexamic Acid in Major Vascular Surgery. A Randomized Placebo-controlled Trial.
Brief Title: Tranexamic Acid in Major Vascular Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Laura Pasin, Medical Doctor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Tranex-AAA/34/OSR
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tranexamic Acid (Experimental): A 500 mg loading dose of tranexamic acid diluted in 100 ml of saline solution will be slowly administered intravenously to patients 20 minutes before surgery, followed by a continuos infusion of 250 mg/h of tranexamic acid from surgical incision until skin closure.
  Interventions: Drug: tranexamic acid diluted in 100 ml of saline solution (loading dose); Drug: tranexamic acid undiluted (continous infusion)
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tranexamic acid diluted in 100 ml of saline solution (loading dose)
  Arms: Tranexamic Acid
Drug: tranexamic acid undiluted (continous infusion)
  Arms: Tranexamic Acid
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether tranexamic acid is effective in reducing intraoperative blood loss and necessity for haemotransfusion in patients undergoing open abdominal aortic aneurysm repair

ELIGIBILITY:
Inclusion Criteria:

* Age > 50
* Able to give written informed consent
* Undergoing open abdominal aortic aneurysm repair

Exclusion Criteria:

* Patients participating in a pharmaceutical clinical trial in the last 3 months
* Urgent/emergent surgery
* Allergy/intolerance to tranexamic acid
* History of seizures
* Acute Venous or Arterial Thrombosis
* Fibrinolytic conditions due to consumption coagulopathy
* Disseminated intravascular coagulation
* Haematuria
* Visual disturbances

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Blood loss (milliliters) | intraoperative (from skin incision to skin closure)

SECONDARY OUTCOMES:
Number of packed blood red cells transfused | hospital stay (an average of one week)
Occurrence of thromboembolic events (of any nature) | 28-days and one year after surgery
Mortality | 28-days and one year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Derived] Monaco F, Nardelli P, Pasin L, Barucco G, Mattioli C, Di Tomasso N, Dalessandro G, Giardina G, Landoni G, Chiesa R, Zangrillo A. Tranexamic acid in open aortic aneurysm surgery: a randomised clinical trial. Br J Anaesth. 2020 Jan;124(1):35-43. doi: 10.1016/j.bja.2019.08.028. Epub 2019 Oct 10. PMID 31607387